CLINICAL TRIAL: NCT00152607
Title: Orthotopic Liver Transplantation Using a Living Donor Into An Adult Recipient
Brief Title: Orthotopic Liver Transplantation Using a Living Donor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10050
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Liver Disease; Liver Neoplasms
Keywords: Liver Transplantation; Living Donors; End Stage Liver Disease
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; End Stage Liver Disease

INTERVENTIONS:
Procedure: donor right hepatic lobectomy

SUMMARY:
The purpose of this study is to:

determine the safety of donor right hepatic lobectomy as a procedure to provide a liver graft for living donor liver transplantation.

study the regeneration of liver tissue by volumetric testing for both donor and recipient.

assess if graft and patient survival with living donor transplantation is comparable to that of cadaveric donor transplantation.

DETAILED DESCRIPTION:
Preoperative Evaluation of Recipients:

Recipients who consent for living donor liver transplantation will have the following measurements performed in addition to those normally performed in their pretransplant workup.

1. Ideal, dry and current body weights.
2. An estimation of the recipient's actual liver volume will be determined by linear CT scanning. Continuous axial-10 mm-thick slices will be obtained following IV contrast. The area of the liver will be electronically outlined on the CT console and then multiplied by the slice thickness. This measurement will be used to assess the accuracy of CT in predicting liver weight and volume by comparing it to the actual volume displacement and weight following hepatectomy.
3. The expected ideal volume of the recipient liver will be calculated from the patient's body weight. Standard liver volume (ml) = 706.2 x (body surface area [m2] + 2.4. Body surface area is calculated from the following formula: BSA = Square root of (Height [inches] x Weight [lbs.]/3131). Example: A recipient who is 5'4" and weighs 121 lbs. has a body surface area of 1.58m2. Thus the estimated ideal liver volume for this recipient is 1120 cc. In order to provide adequate hepatic parenchyma for function they would require 35%-40% of this volume = 392 - 447 cc of liver tissue.

Donor Evaluation:

1. Actual and ideal body weight.
2. History and physical exam.
3. Psychosocial evaluation of the donor will be performed by a social worker for the kidney transplant program. Since he is not affiliated with the liver program, he will be able to objectively assess the potential donor's psychosocial condition. He will continue to see the patient (donor) after the operation while hospitalized and as an outpatient once and then on a prn basis.
4. Evaluations by a donor advocate physician who is not part of the transplant department. The potential donor will be interviewed alone by the physician and allowed to express reservations concerning the procedure in private. The donor advocate physician will review the donor workup in detail to ensure its appropriateness. Should the donor advocate physician indicate that the donor is unsuitable, the donor will be excluded from further evaluation.
5. Donor must be in usual state of health, with normal liver function and no major pre-existing medical conditions.
6. Laboratory testing to rule out concomitant disease that would exclude donation would include the following:

   Blood type and HLA CBC with differential, platelet count Chem 17, SGPT, GGTP, Calcium, Magnesium PT, PTT Pregnancy test for premenopausal women Hepatitis B surface antibody, hepatitis B surface antigen, hepatitis C HIV serology CXR, EKG Cardiac stress test and pulmonary function tests if indicated
7. An estimation of the recipient's right and left lobe size will be determined by linear CT scanning. Continuous axial-10mm-thick slices will be obtained following IV contrast. The area of the liver will be electronically outlined on the CT console and then multiplied by the slice thickness. This measurement will be used to assess the accuracy of CT in predicting liver weight and volume by comparing it to the actual volume displacement and weight following hepatectomy in the donor.
8. Hepatic arteriogram to evaluate the arterial anatomy of the liver.
9. Liver biopsy.
10. Informed consent.

The donor consent is a crucial ethical issue. The donor must be exceptionally well informed concerning the risks of partial hepatectomy. A more difficult element of informed consent, however, is that the donor must make a voluntary choice without coercion. In order to avoid coercion, living donor liver transplants will not be performed in emergency situations. By excluding emergent cases, time to fully consider both the experimental option of living donor transplantation and the standard option of cadaveric donor transplantation will be afforded.

The potential donor will be medically evaluated by an independent (non-study related) physician prior to any consideration of hepatectomy. Karen Kim, M.D., and Sunanda Kane, M.D., both in the section of gastroenterology, will be the donor physician/advocates. We feel that their knowledge of gastroenterology is necessary given the nature of the contemplated surgery, hepatic lobectomy. However, neither of them have affiliations to the liver transplant team, either clinical or research. These physicians will not know the potential recipient's status, will be the final arbiter of the donor's suitability, and will serve as the donor's advocate throughout the transplantation process.

The donor and recipient will both undergo psychosocial evaluation prior to the procedure. This will be to determine psychological suitability for living donor transplantation and to explore personal and family support resources. These interviews will allow both the potential donor and recipient an opportunity to express reluctance to proceed with an individual not directly involved with the transplant procedure. Perhaps the most coercive element for a potential living donor is the perception that it is the expectation of the recipient's family that one should volunteer to donate. This element of coercion can be minimized by allowing the potential donor to discuss any reluctance to donate privately, and apart from their family. They will be reassured that if at any time they do not wish to donate, the recipient will be told only that the donor was not acceptable and the exact reason for this will not be made available. Both the investigators and the donor advocate will perform the process of obtaining informed consent from the donor on two separate occasions not less than one week apart. There will be a thorough discussion of the risks and benefits of the surgery and data will be provided from the short- and long-term follow-up of pediatric donors. These discussions will be with both a transplant hepatologist and surgeon. Once these discussions have taken place, the donor will be given an informed consent form to sign. In seven to ten days, the donor will be approached again regarding liver donation and another consent form will be presented to the donor. After the second consent is signed, it is felt that the donor has met all the physical and emotional requirements for liver donation. If, at the second meeting, the donor requests more time to make an informed consent, this shall be granted. Written consent will also be obtained from the recipient at this time.

Donor Surgical Technique:

1. The donor liver will be partitioned to provide a full right lobe.
2. Intraoperative examination of the liver parenchyma for unsuspected lesions, steatosis will be performed. Intraoperative cholangiography will also be performed to assess the appropriate site of parenchymal transection.
3. Once suitability is confirmed. The appropriate recipient will be brought into the operating room and the hepatectomy begun.
4. During the hepatectomy both the right and left hepatic arteries will be left as long as possible. The portal veins shall be dissected to a level above the confluence of the L & R portal branches.
5. The use of either a right or left lobe will mandate a piggyback technique to be used, as no vena cava will be procured.
6. Arterial anastomosis will be performed with either high-powered loupes or with an operating microscope.

Clearly, information such as actual GWRLW and actual GRBWR will only be available retrospectively (after the donor hepatectomy). The decision to use the donor organ for a living donor liver transplant will be based upon the calculated GWRLW and GRBWR preoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55
2. No current or prior history of heart, lung or other medical problems.
3. No history of liver disease.
4. No history of malignancy, except limited basal cell carcinoma.
5. ABO / HLA compatibility with the recipient.
6. If female and premenopausal, a negative pregnancy test.
7. Related to recipient either by blood or marriage and having a stable, long term, emotional relationship.
8. The donor's body size and volumetric determination of liver mass by abdominal CT scan will indicate whether or not a donor is a suitable candidate for liver donation if the donor meets the other inclusion criteria. Favorable donors for the individual organs will be those with donor graft to recipient body dry weight ratios (GRBWR) of >0.7% and those with a ratio of graft volume to recipient's expected liver volume (GWRLW) of >35%.
9. Satisfactory psychosocial evaluation. -

Exclusion Criteria:

Recipient Exclusion Criteria:

1. Pregnant or nursing females.
2. Patients with significant concomitant infections.
3. Patients who require multiple organ transplants.
4. Significant pulmonary disease. If pulmonary disease is clinically suspected, diagnostic studies will be performed to exclude the presence of pulmonary hypertension (PA systolic pressure >40 mm Hg) or arterial saturation (Po2<60 mmHg, breathing room air).
5. Patients at a higher than average perioperative risk secondary to severe decompensated liver disease or previous surgery (i.e., re-transplantation) or infections.

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2000-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome for donors in this study will be the determination of whether right hepatic lobectomy is a safe procedure for the donor as measured by survival, the incidence of surgical complications, liver function and regeneration studies. | post transplant
The primary outcome for recipients will be the assessment of patient and graft survival. Comparison to results of contemporaneous, non-randomized cadaver donor transplants will be made. | post transplant

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Millis, MD, Principal Investigator — The University of Chicago Hospitals
Locations (1):
- The University of Chicago Hospitals, Chicago, Illinois, United States